CLINICAL TRIAL: NCT02059512
Title: Influence of the Administration of Autologous Bone Marrow Mononuclear Cells for the Duration of Functioning Aorto-coronary Bypass Grafts in the Surgical Treatment of Coronary Heart Disease
Brief Title: Autologous Bone Marrow Mononuclear Cells in the Combined Treatment of Coronary Heart Disease
Acronym: TAMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBK-2901-AMNKM
Record Dates: First submitted 2014-02-01; First posted 2014-02-11 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Ischemic Heart Disease; Bone Marrow Cells; Coronary Artery Bypass Grafting (CABG); Heart Failure, Diastolic
Keywords: ischemic heart disease; bone marrow cells; coronary artery bypass grafting (CABG); reperfusion injury; myocardial dysfunction, diastolic; Heart Failure, Diastolic; transplantation of autologous mononuclear cells; intramyocardial administration; intracoronary administration
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure, Diastolic; Reperfusion Injury; Heart Murmurs

STUDY DESIGN:
Intervention Model Description: Potential participants in this study were all patients admitted for planned coronary artery bypass grafting under extracorporeal circulation and who, according to angiographic examination, had 3 or more stenotic coronary arteries. The final decision on the inclusion of each individual patient in this study was determined taking into account the inclusion criteria. The study was conducted according to the approved protocol as a randomized, blind, placebo controlled.
Who Masked: Investigator
Masking Description: Randomization into three observation groups was carried out according to the table of random numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Intramyocardial administration of autologous bone marrow mononuclear cells during the operation coronary artery bypass grafting 0.2 ml - 10 injection in the zone of blood supply LAD.
  Interventions: Procedure: Group 1
- Group 0 (Placebo Comparator): Intramyocardial administration of 0.9 % NaCl (sodium chloride) 0.2 ml - 10 injection in the zone of blood supply LAD during the operation coronary artery bypass grafting.
  Interventions: Procedure: Group 0
- Group 2 (Active Comparator): Intramyocardial and intracoronary administration of autologous bone marrow mononuclear cells during coronary artery bypass grafting intramyocardial 0.2 ml - 10 injection in the zone of blood supply LAD.
  Interventions: Procedure: Group 2

INTERVENTIONS:
Procedure: Group 1 — Coronary artery bypass grafting with intramyocardial administration of autologous bone marrow mononuclear cells 0.2 ml - 10 injection in the zone of blood supply LAD.
  Other Names: CABG with intramyocardial administration of ABMMC.
  Arms: Group 1
Procedure: Group 0 — Coronary artery bypass grafting with intramyocardial administration of 0.9 % NaCl (sodium chloride) 0.2 ml - 10 injection in the zone of blood supply LAD.
  Other Names: CABG with administration of 0.9 % sodium chlorid.
  Arms: Group 0
Procedure: Group 2 — Coronary artery bypass grafting with intramyocardial and intracoronary administration of autologous bone marrow mononuclear cells intramyocardial administration 0.2 ml - 10 injection in the zone of blood supply LAD.
  Other Names: CABG with intramyocardial and intracoronary administration of ABMMC.
  Arms: Group 2

SUMMARY:
The purpose of this study evaluate the effect of the method of administration of autologous bone marrow mononuclear cells for the duration of of functioning aorto-coronary bypass grafts in the surgical treatment of coronary heart disease, to assess the degree of effectiveness depending on the method of transplantation (intramyocardial, intracoronary, combined).

DETAILED DESCRIPTION:
Additional estimation of safety:

1. Assessment of EuroScore II.
2. Hospital Stay.
3. The duration of stay in the intensive care unit.
4. Restoration of cardiac rhythm at the end of the main stage of operation (defibrillation/ self-recovery).
5. The time of extracorporeal circulation.
6. Time of anoxia.
7. Volume abjointed (drainage) postoperative day 1, day 3
8. Troponin I, CPK-MB, Myoglobin at 1, 3 postoperative days.
9. Hb/ HCT/K+ at the end of cardiopulmonary bypass (CPB) and Hb/ HCT/K+/ ABC at the end of the operation.
10. Assessment of the degree of manifestation of a systemic inflammatory reaction in the postoperative period - leukocytes (Leu), CRP
11. Postoperative complications (hydrothorax, hydropericardium, arrhythmias, resternotomy).
12. Echocardiography at 7-14 days after surgery.

Estimation of efficiency:

1. Evaluation of systolic and diastolic myocardial function. Assessment of myocardial perfusion and metabolism (before and after treatment) - Speckle tracking echocardiography.
2. Patency of grafts within a specified time of treatment (angiography).
3. Dependence and duration of positive clinical effect on the amount of injected cell material.
4. Evaluation of the quality of life (Minnesota questionnaire, Seattle questionnaire, SF- 36 questionnaire).
5. All-cause Mortality Associated With the Progression of Basic
6. Disease.Dynamics of the functional class of angina.
7. Dynamics of the functional class of heart failure.
8. Dynamics of test data with a 6-minute walk.

Predicting the results of treatment (the effect of a number of parameters):

1. Age.
2. Gender.
3. The body mass index.
4. Diabetes.
5. Smoking.
6. Family history of cardiovascular events.
7. Duration of ischemic heart disease.
8. Serum total cholesterol (+ fractions).
9. Leukocytosis and CRP level (initial level and rate of decrease in the postoperative period).
10. The level of creatinine.
11. The presence / absence of extracardiac arteriopathy.
12. The intramyocardial or intracoronary injection of BM-MNCs.
13. Assessment of the bone marrow: the number of nucleated cells, CD34 +, CD133 +.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 80 years
* Patients with angina pectoris III-IV functional class
* According to angiographic examination, the presence of 3 or more stenotic coronary arteries
* Aorto-coronary bypass surgery under cardiopulmonary bypass
* Patients signed informed consent

Exclusion Criteria:

* Intolerance of heparin and HES.
* Hypothyroidism and hyperthyroidism.
* Associated pathology with a projected lifespan limitation to 3 years.
* infection diseases
* Simultaneous participation in another study.
* Pregnancy.
* Severe mental disorder.
* Refusal of a patient to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Komok, Ph.D, Principal Investigator — First Pavlov State Medical University of St. Petersburg.
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Komok V.V., Bunenkov N.S., Beliy S.A., Pizin V.M., Kondratev V.M., Dulaev А.V., Lukashenko V.I., Kobak A.E., Maksimova T.S., Sergienko I.P., Parusova E.V., Smirnova L.A., Babenko E.V., Afanasev B.V., Nemkov A.S., Khubulava G.G. Assessment of safety of additional transplantation of autologous bone marrow mononuclear cells in the combined treatment of coronary heart disease. Results from a randomized, blind, placebo-controlled trial (TAMIS). Russian Journal of Transplantology and Artificial Organs. 2019;21(2):112-120. (In Russ.) https://doi.org/10.15825/1995-1191-2019-2-112-120
- [Background] Komok V.V., Bunenkov N.S., Beliy S.A., Pizin V.M., Kondratev V.M., Dulaev A.V., Kobak A.E., Maksimova T.S., Sergienko I.P., Parusova E.V., Smirnova L.A., Babenko E.V., Afanasev B.V., Nemkov A.S., Khubulava G.G. Evaluation of the effectiveness of combined treatment of coronary heart disease - coronary artery bypass grafting, transplantation of autologous bone marrow mononuclear cells: a randomized, double-blind, placebo-controlled study. Russian Journal of Transplantology and Artificial Organs. 2019;21(4):54-66. https://doi.org/10.15825/1995-1191-2019-4-54-66
- See also: Assessment of safety of additional transplantation of autologous bone marrow mononuclear cells in the combined treatment of coronary heart disease. Results from a randomized, blind, placebo-controlled trial (TAMIS). — https://journal.transpl.ru/vtio/article/view/1027
- See also: Evaluation of the effectiveness of combined treatment of coronary heart disease - coronary artery bypass grafting, transplantation of autologous bone marrow mononuclear cells: a randomized, double-blind, placebo-controlled study. — https://journal.transpl.ru/vtio/article/view/1106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants in the study were all patients referred to the clinic for surgical treatment of coronary artery disease.
Pre-assignment Details: The study included patients admitted for routine coronary artery bypass grafting under cardiopulmonary bypass, and having, according to the angiographic studies, 3 or more of stenosed coronary arteries. Patients met the inclusion criteria and signed an informed voluntary consent.
Groups:
- Intramyocardial Administration 0.9 % NaCl (Sodium Chloride) - Group 0: Сoronary artery bypass grafting with intramyocardial administration of 0.9 % NaCl (sodium chloride) 0.2 ml - 10 injection in the zone of blood supply LAD.
- Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1: Сoronary artery bypass grafting with intramyocardial administration of autologous bone marrow stem cells 0.2 ml - 10 injection in the zone of blood supply LAD.
- Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2: Сoronary artery bypass grafting with intramyocardial (0.2 ml - 10 injection in the zone of blood supply LAD) and intracoronary administration of autologous bone marrow stem cells.
Period: Overall Study
Arm/Group | Intramyocardial Administration 0.9 % NaCl (Sodium Chloride) - Group 0 | Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1 | Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2
Started | 46 | 34 | 37
Completed | 37 | 25 | 23
Not Completed | 9 | 9 | 14

BASELINE CHARACTERISTICS:
Population: The study included patients admitted for coronary artery bypass grafting. Patients met the inclusion criteria and signed an informed consent.
  In the "results" section, data are provided for repeated examinations of patients.
Groups:
- Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1: Сoronary artery bypass grafting with intramyocardial administration of autologous bone marrow mononuclear cells 0.2 ml - 10 injection in the zone of blood supply LAD.
- Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2: Сoronary artery bypass grafting with intramyocardial ( 0.2 ml - 10 injection in the zone of blood supply LAD) and intracoronary administration of autologous bone marrow mononuclear cells.
- Total: Total of all reporting groups
Arm/Group | Intramyocardial Administration 0.9 % NaCl (Sodium Chloride) - Group 0 | Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1 | Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2 | Total
Number analyzed (Participants) | 37 | 25 | 23 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 18 | 20 | 67
  >=65 years | 8 | 7 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 61.7 (6.8) | 59.5 (5.4) | 60.9 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender sign: Female, Male Population: The analysis of the final statistics was made at the time the studies were completed.
  Participants
    Female | 6 | 4 | 3 | 13
    Male | 31 | 21 | 20 | 72
Region of Enrollment [Number; unit: participants] — North-West Russia:Novgorod region, Leningrad region, Pskov region.
  participants
    Russia | 37 | 25 | 23 | 85
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI (body mass index) = weit (kg)/(height (m))^2 Norm (18.5-25); 1-overweight (25-30); I degree of obesity (30-35); II degree of obesity (35-40); III degree of obesity (40 and>).
  kg/m^2 | 28.6 (3.59) | 28.05 (4.46) | 28.09 (3.57) | 28.3 (3.4)
Diabetes [Count of Participants; unit: Participants] — According to laboratory data - compensated (diet, drug therapy, insulin).
  Participants | 6 | 5 | 4 | 15
Hypertonic desease (stage). [Count of Participants; unit: Participants] — 2 stage - Blood pressure ranges from 160/100 to 179/109 mm Hg. There are signs of damage to the heart, retina and kidneys, which can only be detected by instrumental or laboratory examination methods. There are no subjective symptoms of their defeat.
  3 stage - Blood pressure is 180/110 mm Hg. and higher. There are objective signs and subjective symptoms of the heart, the brain, retina, kidney, or blood vessels.
  Stage 2 is associated with a lower risk of adverse cardiovascular events.
  Participants
    2 stage | 1 | 0 | 0 | 1
    3 stage | 36 | 25 | 23 | 84
Arterial hypertension (degree) [Count of Participants; unit: Participants] — 1. degree - Blood pressure ranges from 140/90 to 159/99 mm. Hg
  2. degree - Blood pressure ranges from 160/100 to 179/109 mm Hg.
  3. degree - Blood pressure is 180/110 mm Hg. and higher.
  Degree 1 and 2 is associated with a lower risk of adverse cardiovascular events.
  Participants
    No | 2 | 3 | 2 | 7
    1 degree | 6 | 5 | 5 | 16
    2 degree | 14 | 11 | 7 | 32
    3 degree | 15 | 6 | 9 | 30
Peripheral arteriopathy. [Count of Participants; unit: Participants] — The presence of peripheral arteriopathy (hemodynamically significant stenosis in the carotid arteries, arteries of the lower extremities).
  According to ultrasound, angiographic research methods: carotid arteries, lower limb arteries.
  Participants | 11 | 4 | 6 | 21
Acute myocardial infarction transferred in history (number). [Count of Participants; unit: Participants]
  1 acute myocardial infarctions | 14 | 17 | 9 | 40
  2 acute myocardial infarctions | 4 | 3 | 6 | 13
  3 acute myocardial infarctions | 2 | 1 | 1 | 4
Smoking. [Count of Participants; unit: Participants] — Active smoking at the time of hospitalization for routine CABG.
  Participants | 7 | 2 | 4 | 13
Family history of cardiovascular disease. [Count of Participants; unit: Participants] — Family history of cardiovascular disease: hypertension, arterial hypertension, AMI, stroke, the presence of peripheral arteriopathy requiring medical intervention.
  Participants | 19 | 11 | 10 | 40
Debut of ischemic heart disease (months). [Mean (Standard Deviation); unit: months] | 71.9 (70.9) | 62.9 (79.2) | 76.9 (59.4) | 69.3 (60.3)
Debut of ischemic heart disease. [Count of Participants; unit: Participants]
  Debut of ischemic heart disease up to 5 years | 23 | 16 | 12 | 51
  Debut of ischemic heart disease 6-10 years | 8 | 4 | 8 | 20
  Debut of ischemic heart disease over 10 years | 6 | 5 | 3 | 14
Angina pectoris (functional class). [Count of Participants; unit: Participants] — 2 functional class - Pain attacks when walking more than 500 meters, when climbing stairs more than one floor.
  3 functional class. Attacks when walking on level ground at 100-500 meters, when climbing stairs one floor.
  4 functional class. Seizures when walking on level ground at a distance of less than 100 meters, and when at rest.
  Painless myocardial ischemia is characterized by changes in myocardial blood supply without pain.
  The lower the functional class of angina pectoris, the better the quality of life.
  Participants
    2 functional class | 1 | 0 | 0 | 1
    3 functional class | 32 | 23 | 21 | 76
    4 functional class | 3 | 2 | 1 | 6
    painless ischemia | 1 | 0 | 1 | 2
Heart failure (functional class NYHA). [Count of Participants; unit: Participants] — 1. functional class - There is no limitation of a person's physical activity, shortness of breath manifests itself when going above the third floor.
  2. functional class - slight limitation of activity, palpitations, shortness of breath, fatigue occur during normal physical activity and more.
  3. functional class - Symptoms occur with the smallest physical activity, resulting in a significant decrease in activity. At rest, clinical manifestations are not observed.
  The smaller the functional class, the better the quality of human life.
  Participants
    1 functional class | 5 | 1 | 2 | 8
    2 functional class | 29 | 24 | 21 | 74
    3 functional class | 3 | 0 | 0 | 3
Total holesterol (mmol/l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 4.49 (1.08) | 4.5 (1.24) | 4.6 (1.49) | 4.5 (1.1)
Very loud density lipoprotein (mmol/l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 0.96 (0.35) | 0.94 (0.5) | 0.77 (0.3) | 0.95 (0.31)
High density lipoproteins (mmol/l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 2.7 (0.89) | 2.58 (1.05) | 2.7 (1.26) | 2.6 (1.1)
Loud density lipoproteins (mmol/l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 0.98 (0.31) | 1.16 (0.37) | 1.13 (0.29) | 1.1 (0.3)
Triglyceride (mmol/l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 2.04 (0.68) | 1.69 (0.72) | 1.63 (0.62) | 1.9 (0.65)
Atherogenic coefficient. [Mean (Standard Deviation); unit: ratio] — The data at the time of hospitalization for routine CABG. Atherogenic Coefficient (AC) is a predictor of the risk of coronary artery disease and is calculated as {(Total Cholesterol - HDLc)/HDLc}.
  ratio | 4.07 (1.32) | 3.27 (1.9) | 4.5 (5.2) | 4.08 (2.1)
Creatinine (mmol / l). [Mean (Standard Deviation); unit: mmol/l] — The data at the time of hospitalization for routine CABG.
  mmol/l | 0.09 (0.02) | 0.09 (0.02) | 0.08 (0.02) | 0.09 (0.02)
C-reactive protein (mg/l). [Mean (Standard Deviation); unit: mg/l] — The data at the time of hospitalization for routine CABG.
  mg/l | 5.9 (11.07) | 2.56 (1.96) | 5.3 (5.38) | 4.9 (6.8)
Glomerular filtration rate (ml/min/1.73 m^2) (assessment of renal function). [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — The CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration Formula):scale was used to assess renal function. The degree of renal dysfunction was assessed according to https://www.kidney.org/professionals/explore-your-knowledge/how-to-classify-ckd The standards are as follows: Category G1 ≥90 ml/min/1.73 m^2 (Normal or high); G2 - 60-89 ml/min/1.73 m^2 (Mildly decreased); G3a - 45-59 ml/min/1.73 m^2 (Mildly to moderately decreased); G3b - 30-44 ml/min/1.73 m^2 (Moderately to severely decreased); G4 15-29 ml/min/1.73 m^2 (Severely decreased); G 5 <15 ml/min/1.73 m^2 (Kidney failure).
  ml/min/1.73 m^2 | 79.89 (15.8) | 77.6 (16.03) | 84.2 (17.26) | 77.9 (16.8)
EuroScore II [Mean (Standard Deviation); unit: percentage of risk] — EuroScoreII is designed to assess the risk of adverse outcome in coronary artery bypass grafting. Assessment factors: age, gender, serum creatinine, extracardiac artery disease, chronic lung disease, severe neurological disorders, previous cardiac surgery, previous myocardial infarction, left ventricular dysfunction, diabetes mellitus, pulmonary hypertension, grade IV angina pectoris, active endocarditis, unstable angina pectoris, surgery, critical condition of the patient before surgery, type of surgery. The higher the score, the higher the risk of an adverse outcome.
  percentage of risk | 1.3 (0.68) | 1.07 (0.47) | 1.02 (0.4) | 1.15 (0.5)
SYNTAX Score [Mean (Standard Deviation); unit: units on a scale] — The SYNTAX Score Calculator is a scale developed in connection with the SYNTAX study The scale includes an assessment of the nature of the anatomical structure and atherosclerotic lesions of the coronary arteries. Each factor has a certain score. Based on the summation of the scores, the risk stratification is assessed. The following risk groups have been identified. Low-risk group with a score of 0-22, medium-risk group 23-32 points, high-risk group> 32 points. http://www.syntaxscore.com/calculator/syntaxscore/frameset.htm
  units on a scale | 26.7 (7.0) | 26.8 (6.0) | 26.4 (7.3) | 26.7 (6.4)
Nitrates. [Count of Participants; unit: Participants] — Number participants who were receiving Nitrates treatment. Basic therapy for hospitalization for planned CABG.
  Participants | 21 | 11 | 10 | 42
Diuretics. [Count of Participants; unit: Participants] — Number participants who were receiving Diuretics treatment. Basic therapy for hospitalization for planned CABG.
  Participants | 5 | 10 | 3 | 18
Angiotensin converting enzyme inhibitors. [Count of Participants; unit: Participants] — Number participants who were receiving Angiotensin converting enzyme inhibitors treatment. Basic therapy for hospitalization for planned CABG.
  Participants | 18 | 9 | 16 | 43
Angiotensin receptor antagonists. [Count of Participants; unit: Participants] — Number participants who were receiving Angiotensin receptor antagonists treatment.Basic therapy for hospitalization for planned CABG.
  Participants | 5 | 3 | 4 | 12
β-blockers. [Count of Participants; unit: Participants] — Number participants who were receiving β-blockers treatment.Basic therapy for hospitalization for planned CABG.
  Participants | 35 | 20 | 23 | 78
Antagonists СА - calcium tubules antagonists. [Count of Participants; unit: Participants] — Number participants who were receiving Antagonists СА - calcium tubules antagonists treatment. Basic therapy for hospitalization for planned CABG.
  Participants | 5 | 6 | 4 | 15
Antiplatelet agents. [Count of Participants; unit: Participants] — Number participants who were receiving Antiplatelet agent treatment.Basic therapy for hospitalization for planned CABG.
  Participants | 18 | 12 | 9 | 39
Anticoagulants. [Count of Participants; unit: Participants] — Number participants who were receiving Anticoagulants treatment.Basic therapy for hospitalization for planned CABG.
  Participants | 6 | 0 | 2 | 8
Statins. [Count of Participants; unit: Participants] — Number participants who were receiving Statins treatment. Basic therapy for hospitalization for planned CABG.
  Participants | 27 | 16 | 15 | 58
Echocardiography - 1. Lvd ind. Lvs ind. LAind. [Mean (Standard Deviation); unit: mm/ m^2] — The data at the time of hospitalization for routine CABG. Indicators of size of the left chambers of the heart. Lvd ind. - left ventricular end-diastolic size index; Lvs ind. - left ventricular end-systolic size index; LA ind. - left atrial index.
  The greater figure (size of the left ventricle - index), worse the prognosis of adverse outcome.The index is used as an indicator of the payment to obtain a more reliable result (taking into account individual characteristics of each patient).
  index - size of the left ventricle/ body mass index (kg / m^2).
  mm/ m^2
    Lvd ind. | 2.7 (0.39) | 2.98 (0.5) | 2.8 (0.2) | 2.8 (0.36)
    Lvs ind. | 1.8 (0.42) | 2.1 (0.5) | 1.9 (0.4) | 1.9 (0.44)
    LAind. | 2.1 (0.3) | 2.2 (0.3) | 2.1 (0.2) | 2.2 (0.27)
Echocardiography - 2. LVEDV MOD BP ind. LVESV MOD BP ind. [Mean (Standard Deviation); unit: ml/ m^2] — The data at the time of hospitalization for routine CABG. Volume indices of left heart chambers.
  LVEDV MOD BP ind. - left ventricular end-diastolic volume index. LVESV MOD BP ind. - left ventricular end-systolic volume index.
  The greater figure (size of the left ventricle - index), worse the prognosis of adverse outcome.The index is used as an indicator of the payment to obtain a more reliable result (taking into account individual characteristics of each patient).
  index - size of the left ventricle/ body mass index (kg / m^2).
  ml/ m^2
    LVEDV MOD BP ind. | 62.4 (20.7) | 73 (36.1) | 73.2 (29.9) | 62.7 (28.9)
    LVESV MOD BP ind. | 23.6 (14.8) | 32.4 (27.9) | 31.9 (22.3) | 27.9 (21.7)
Echocardiography - 3. LVEF (Simpson) - left ventricular ejection fraction. [Mean (Standard Deviation); unit: percent] — The data at the time of hospitalization for routine CABG. Assessment of the contractility of the left ventricular myocardium (systolic function)
  percent | 62.1 (7.4) | 56.6 (10.2) | 59.3 (11.1) | 59.8 (9.6)
Echocardiography - 4. Left ventricular diastolic function - 1. [Mean (Standard Deviation); unit: m/sec] — Evaluation of left ventricular diastolic function (echocardiography). The peak velocity E reflects the pressure gradient between the LA and LV in early diastole, and it is affected by preload and disturbance LV relaxation The speed of peak A, which forms at the end diastole, influences LV compliance and contractility left atrium.
  m/sec
    Peak E of transmitral flow | 0.7 (0.2) | 0.6 (0.1) | 0.7 (0.2) | 0.7 (0.2)
    Peak A of transmitral flow | 0.8 (0.2) | 0.8 (0.2) | 0.7 (0.2) | 0.7 (0.2)
Echocardiography - 5. Left ventricular diastolic function - 2 (E/A). [Mean (Standard Deviation); unit: ratio] — The ratio of the transmitral flow, wave E (ejection wave / left ventricular contraction) to wave A (ejection wave / left atrial contraction). The norm is 0.75-1.5 Less than 0.75 violation of relaxation, more than 1.5 restrictive type of diastolic dysfunction.
  ratio | 0.9 (0.4) | 0.9 (0.5) | 0.9 (0.5) | 0.9 (0.47)
Echocardiography - 6. Left ventricular diastolic function - 3 (DT, IVRT). [Mean (Standard Deviation); unit: ms.] — Assessment of left ventricular diastolic function. The data at the time of hospitalization for routine CABG. DT (Half-time of wave E). The DT time index reflects the relaxation process LV, LV diastolic pressure after mitral valve opening, and LV compliance. 150-200 ms - normal; > 200 ms - violation of relaxation; 150-200 ms - pseudonormal type of left ventricular filling; <150 ms - restrictive type of diastolic dysfunction IVRT (time of isovolumic relaxation of the left ventricl.) <100 ms - normal; > 100 ms - violation of relaxation
  ms.
    DT (Half-time of wave E) | 253 (52.7) | 257.6 (46.3) | 252.3 (55.1) | 254.7 (51.4)
    IVRT (time of isovolumic relaxation of the left ventriclar) | 103.4 (11.1) | 106 (9.8) | 105.3 (13.9) | 104.7 (11.6)
Echocardiography - 7. LVmass/ BSA (g/m^2) [Mean (Standard Deviation); unit: g/m^2] — left ventricular mass (LVmass)/ body surface area (BSA) = left ventricular mass index (g/m^2).
  Men - normal - 115 g / m^2 Women - normal - 95 g / m^2
  g/m^2 | 119.1 (29) | 152.8 (48) | 134.04 (32) | 135.3 (36.3)
Echocardiography - 8. RWT - relative wall thickness of the left ventricle. [Mean (Standard Deviation); unit: ratio] — Calculated by the formula left ventricular posterior wall thickness + interventricular septal thickness / left ventricular end-diastolic size.
  RWT more 0.42 - concentric hypertrophy of the left ventricular myocardium. RWT less or equal 0.42 - eccentric left ventricular myocardial hypertrophy.
  ratio | 0.44 (0.07) | 0.4 (0.07) | 0.4 (0.06) | 0.43 (0.07)
Echocardiography - 9. Mitral regurgitation. [Count of Participants; unit: Participants] — The data at the time of hospitalization for routine CABG. Evaluation of the degree of Mitral regurgitation by echocardiography data.
  Assessment of the degree by the ratio of the area of the regurgitation stream to the area of the left atrium:
  Grade 1 (easy) - less than 20% Grade 2 (moderate) - 20-40% Grade 3 (severe) - more than 40% Valve insufficiency is absent in the norm. 2 degree of failure - requires dynamic observation. 3-4 degree of failure requires further examination, the decision of the HeartTeam about the need for surgical correction.
  Participants
    Not | 16 | 8 | 6 | 30
    1 degree Mitral regurgitation. | 19 | 13 | 13 | 45
    2 degree Mitral regurgitation. | 2 | 3 | 3 | 8
    3 degree Mitral regurgitation. | 0 | 1 | 1 | 2
Echocardiography - 10. Tricuspid regurgitation. [Number; unit: participants] — Criteria tricuspid regurgitation. Grade1-central jet area regurgitation<5.0 cm^2, Vena contracta is minimal.Grade2-The area of central jet area regurgitation is 5.0-10cm^2, Vena contracta is <0.7cm. Grade 3-central jet area regurgitation>10cm^2, Vena contracta>0.7cm Additional criterion - retrograde movement of blood in the hepatic vein during systole. Valve insufficiency is absent in the norm. 2degree of failure-requires dynamic observation. 3-4degree of failure requires further examination, the decision of the HeartTeam abCriteria tricuspid insufficiency out the need for surgical correction.
  participants
    Not | 25 | 22 | 19 | 66
    1 degreeTricuspid regurgitation | 12 | 3 | 4 | 19
    2 degreeTricuspid regurgitation | 0 | 0 | 0 | 0
    3 degreeTricuspid regurgitation | 0 | 0 | 0 | 0
Echocardiography - 11. Aortic regurgitation. [Number; unit: participants] — Evaluation of the degree of Aortic regurgitation by echocardiography data.
  Ultrasound criteria for the significance of aortic valve insufficiency are determined by the time of the half-decay of the diastolic gradient of the aortic regurgitation flow:
  1 stage more than 400 ms; 2 stage 250-400 ms; 3 degree less than 250ms Valve insufficiency is absent in the norm. 2 degree of failure - requires dynamic observation. 3-4 degree of failure requires further examination, the decision of the HeartTeam about the need for surgical correction.
  participants
    Not | 25 | 23 | 22 | 70
    1 degree Aortic regurgitation. | 11 | 2 | 1 | 14
    2 degree Aortic regurgitation. | 1 | 0 | 0 | 1
    3 degree Aortic regurgitation. | 0 | 0 | 0 | 0
Echocardiography - 12. Signs of myocardial remodeling. [Count of Participants; unit: Participants] — The data at the time of hospitalization for routine CABG
  Participants
    Left ventricular diastolic function/: Yes | 19 | 17 | 16 | 52
    Left ventricular diastolic function/: Not | 18 | 8 | 7 | 33
    Left ventricular aneurysm.: Yes | 2 | 4 | 3 | 9
    Left ventricular aneurysm.: Not | 35 | 21 | 20 | 76
    Change in local kinetics.: Yes | 23 | 11 | 12 | 46
    Change in local kinetics.: Not | 14 | 14 | 11 | 39

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Initial Risk of Surgery (EuroScore II).
Description: EuroScoreII is intended to assess the risk of adverse outcome of coronary artery bypass grafting. Assessment factors: age, sex, serum creatinine, extracardiac artery disease, chronic lung disease, severe neurological disorders, previous cardiac surgery, previous myocardial infarction, left ventricular dysfunction, diabetes mellitus, pulmonary hypertension, IV class of angina severity, active endocarditis, unstable angina, surgery, critical condition of the patient before surgery, type of surgery. The higher the percentage, the higher the risk of surgery.
Time Frame: Before CABG surgery at baseline.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Group 0: Сoronary artery bypass grafting with intramyocardial administration of 0.9 % NaCl (sodium chloride) 0.2 ml - 10 injection in the zone of blood supply LAD.
- Group 1: Сoronary artery bypass grafting with intramyocardial administration of autologous bone marrow stem cells 0.2 ml - 10 injection in the zone of blood supply LAD.
- Group 2: Сoronary artery bypass grafting with intramyocardial (0.2 ml - 10 injection in the zone of blood supply LAD) and intracoronary administration of autologous bone marrow stem cells.
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
percent | 1.3 (0.68) | 1.07 (0.47) | 1.02 (0.4)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.24, Kruskal-Wallis

2. Primary Outcome: Length of Hospital Stay. Length of Stay in the Intensive Care Unit.
Description: The results were obtained from the analysis of primary data.
Time Frame: Primary hospitalization for planned CABG.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Group 0: Сoronary artery bypass grafting with intramyocardial administration of 0.9 % NaCl (sodium chloride) 0.2 ml - 10 injection in the zone of blood supply LAD.
  Сontrol group.
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
days
  Hospital Stay | 36.8 (11.2) | 32.8 (13.9) | 38.4 (15.2)
  Days in the intensive care unite | 3.9 (2.2) | 3.1 (1.7) | 3.3 (1.8)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Length of hospital stay; Test type: Superiority; p = 0.1, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Length of stay in the intensive care unit; Test type: Superiority; p = 0.1, Kruskal-Wallis

3. Primary Outcome: The Severity of the Systemic Inflammatory Response in the Postoperative Period (Leukocytosis).
Description: Assessment of the severity of the systemic inflammatory response during hospital stay after surgery. Assessment of the level of inflammation by the severity of an increase in leukocytes (leukocytosis).
  Leukocytosis - an increase in the number of leukocytes per unit volume of blood. The norm of leukocytes in the blood is 5.5-8.810^9 /l. For adults, leukocytosis is considered to be an increase in the number of leukocytes in the blood of more than 9.0*10^9 / l In the statistical analysis, the grouping of indicators in the indicated intervals was used, in view of the individual characteristics of the course of the postoperative period in each case.
Time Frame: The parameters were evaluated initially at baseline in the postoperative period - an interval of 0-6 hours, 12-18 hours, 18-24 hours, 48 hours, 72 hours, 96 hours, 7 days and 14 days.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: x10^9 cells/L"
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
x10^9 cells/L"
  Leu (leukocytes) / initially | 8.3 (2.2) | 6.5 (1.5) | 7.3 (2.04)
  Leu / in the postoperative period - an interval of 0-6 hours | 13.9 (6.3) | 14.1 (1.9) | 16.2 (5.4)
  Leu / in the postoperative period - an interval of 12-18 hours | 13.9 (3.99) | 14.7 (5.9) | 13.3 (3.7)
  Leu / in the postoperative period - an interval of 18-24 hours | 13.08 (2.4) | 15.4 (2.4) | 16.99 (3.9)
  Leu / in the postoperative period 48 hours | 13.8 (5.5) | 14.8 (2.2) | 13.3 (3.97)
  Leu / in the postoperative period 72 hours | 11.3 (4.1) | 9.4 (1.6) | 11.4 (1.9)
  Leu / in the postoperative period 96 hours | 10.1 (2.7) | 8.7 (2.6) | 10.4 (1.99)
  Leu / in the postoperative period 7 days | 11.9 (5.9) | 9.5 (2.3) | 10.4 (3.2)
  Leu / in the postoperative period 14 days | 8.8 (1.6) | 8.8 (1.7) | 10.4 (3.06)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 0-6 hours of the postoperative period; Test type: Superiority; p = 0.8, Kruskal-Wallis
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 12-18 hours of the postoperative period; Test type: Superiority; p = 0.9, Kruskal-Wallis
Statistical Analysis 4: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 18-24 hours of the postoperative period; Test type: Superiority; p = 0.2, Kruskal-Wallis
Statistical Analysis 5: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 48 hours of the postoperative period; Test type: Superiority; p = 0.5, Kruskal-Wallis
Statistical Analysis 6: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 72 hours of the postoperative period; Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 7: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 96 hours of the postoperative period/; Test type: Superiority; p = 0.6, Kruskal-Wallis
Statistical Analysis 8: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 7 days of the postoperative period; Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 9: Comparison: Group 0 vs Group 1 vs Group 2; Analysis of leukocytes 14 days of the postoperative period; Test type: Superiority; p = 0.5, Kruskal-Wallis

4. Primary Outcome: Assessment of the Degree of General Inflammatory Response (C-reactive Protein (CRP)),
Description: Results of dynamic control of laboratory parameters of CRP. C-reactive protein. This fraction of plasma proteins increases in the presence of an inflammatory process in the body. It is synthesized in response to the ingestion of toxins of pathological microorganisms into the bloodstream and neutralizes them by binding them. In addition, it appears when the body's own cells are destroyed in the event of necrosis, tumor disintegration or extensive trauma, inactivating the resulting products. In addition to eliminating toxins, CRP triggers a cascade of immune responses aimed at eliminating pathologically altered structures.
  Normally absent (or less than 0.4 mg / l). In the statistical analysis, the grouping of indicators in the indicated intervals was used, in view of the individual characteristics of the course of the postoperative period in each case.
Time Frame: Initial data, control point in the interval 4-6 days of the postoperative period, control point in the interval 12-14 days of the postoperative period.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mg/l
  CRP initially/ mg / l | 4.4 (6.05) | 3.05 (2) | 5.1 (5.1)
  CRP control point in the interval 4-6 days of the postoperative period/ mg/l | 80.2 (38) | 85.9 (51.8) | 121.1 (76.3)
  CRP control point in the interval 12-14 days of the postoperative period/ mg/l | 24.6 (13.8) | 25.9 (20.9) | 24.4 (15.6)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; CRP initially; Test type: Superiority; p = 0.1, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; CRP postoperative 4-6 days; Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; CRP postoperative 12-14 days; Test type: Superiority; p = 0.99, Kruskal-Wallis

5. Primary Outcome: The Volume of Discharge Through the Drains in the Early Postoperative Period.
Description: A daily assessment of the discharge by drainage before removal was carried out. It was carried out to assess the possible development of an excessive inflammatory reaction (polyserositis phenomena) in response to the transplantation of autologous bone marrow mononuclear cells.
Time Frame: Evaluation of these data - for the time spent in the intensive care unit before removing the drains.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
milliliters
  The volume of discharge through the drains on the first day after surgery. | 541.2 (47.9) | 424 (95.7) | 410 (59.4)
  The volume of discharge through the drains on the second day after the operation. | 189.7 (27.1) | 152 (54.2) | 195.4 (33.6)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; The volume of discharge through the drains on the first day after surgery; Test type: Superiority; p = 0.2, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; The volume of discharge through the drains on the second day after the operation; Test type: Superiority; p = 0.3, RepeatedMeasures ANOVA

6. Primary Outcome: Dynamics of Markers of Myocardial Damage (Troponin I, Myoglobin).
Description: Assessment of the severity of the period of ischemia / reperfusion. And the effect of autologous bone marrow mononuclear cells transplantation on these indicators.
Time Frame: 1 and 3 days of the postoperative period.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: mcg / l
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mcg / l
  Troponin I (postoperative day 1)/mcg / l | 12.05 (18.9) | 5.7 (5.8) | 2.9 (2.3)
  Troponin I (postoperative day 3)/mcg / l | 19.6 (31.9) | 3.08 (3.7) | 1.9 (1.3)
  Myoglobin postoperative day 1/mcg / l/ | 522.8 (711.6) | 385.6 (221.7) | 757.2 (1146.8)
  Myoglobin postoperative day 3/mcg / l | 92.5 (1094.8) | 71.4 (41.4) | 70.4 (148.4)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Troponin I postoperative day 1; Test type: Superiority; p = 0.6, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Troponin I postoperative day 3; Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; Myoglobin postoperative day 1; Test type: Superiority; p = 0.8, Kruskal-Wallis
Statistical Analysis 4: Comparison: Group 0 vs Group 1 vs Group 2; Myoglobin postoperative day 3; Test type: Superiority; p = 0.7, Kruskal-Wallis

7. Primary Outcome: Dynamics of Markers of Myocardial Damage (Creatine Phosphokinase Fraction MB (CPK-MB)).
Description: as for outcome 6
Time Frame: 1 and 3 days of the postoperative period.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
U/l
  CPK-MB postoperative day 1/ U/l | 62.3 (1024) | 63.02 (79.2) | 78.6 (136.8)
  CPK-MB postoperative day 3/ U/l | 35.4 (84.7) | 9.5 (9.3) | 4.6 (1.9)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; CPK-MB postoperative day 1; Test type: Superiority; p = 0.7, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; CPK-MB postoperative day 3; Test type: Superiority; p = 0.8, Kruskal-Wallis

8. Primary Outcome: Intraoperative Assessment of Homeostasis (Hemoglobin (Hb).
Description: These parameters were evaluated at the end of the cardiopulmonary bypass and at the end of the surgery. The interval between indicators is on average from 60 to 120 minutes.
Time Frame: Intraoperative data.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
g/l
  Hb intraoperatively before turning off the cardiopulmonary bypass (CPB). | 74.05 (12.2) | 73.4 (8.08) | 75.8 (14.5)
  Hb at the end of the operation. | 91.3 (16.09) | 91.5 (8.6) | 86.7 (11.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Hb intraoperatively before turning off the cardiopulmonary bypass(CPB); Test type: Superiority; p = 1.0, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Hb at the end of the operation; Test type: Superiority; p = 0.4, Kruskal-Wallis

9. Primary Outcome: Intraoperative Assessment of Homeostasis (Hematocrit (HCT)).
Description: as for outcome 8
Time Frame: Intraoperative data.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
percent
  HCT intraoperatively before turning off the cardiopulmonary bypass(CPB). | 23.4 (4.2) | 22.2 (1.9) | 23.2 (3.9)
  HCT at the end of the operation. | 29.3 (5.2) | 27.8 (3.2) | 25.7 (3.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; HCT intraoperatively before turning off the cardiopulmonary bypass (CPB); Test type: Superiority; p = 0.8, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; HCT at the end of the operation; Test type: Superiority; p = 0.3, Kruskal-Wallis

10. Primary Outcome: Intraoperative Assessment of Homeostasis (К+).
Description: as for outcome 8
Time Frame: Intraoperative data.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mmol/l
  K+ intraoperatively before turning off the cardiopulmonary bypass(CPB). | 5.01 (0.59) | 5.4 (0.9) | 4.7 (0.9)
  K+ at the end of the operation. | 3.9 (0.4) | 4.5 (0.6) | 3.9 (0.5)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; K+ intraoperatively before turning off the cardiopulmonary bypass (CPB); Test type: Superiority; p = 0.4, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; K+ at the end of the operation; Test type: Superiority; p = 0.1, Kruskal-Wallis

11. Primary Outcome: Cardiopulmonary Bypass Time.
Time Frame: Intraoperative data.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
minutes | 135 (31.6) | 122.8 (19.7) | 144 (29.2)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.1, Kruskal-Wallis

12. Primary Outcome: Time of Aortic Clamping (Anoxia).
Description: Estimation of the time from the moment the clamp is applied to the aorta (complete clamping of the aorta) to the removal of the clamp from the aorta.
Time Frame: Intraoperative data.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
minutes | 75.8 (17.6) | 73.8 (22.3) | 84 (18.8)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.1, Kruskal-Wallis

13. Primary Outcome: Assessment of Complications in the Postoperative Period. Additional Estimation of Safety.
Description: The presence of complications in the postoperative period (Hydrothorax, Hydropericardium, Cardiac arrhythmias - atrial fibrillation / atrial flutter).
Time Frame: Postoperative period.
Population: The data of all patients initially included in the study were analyzed.
Measure: Number; unit: participants
Arm/Group | Group 0. | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
participants
  Hydrothorax / postoperative period | 3 | 4 | 3
  Hydropericardium / postoperative period | 0 | 1 | 2
  Resternotomy / postoperative period | 1 | 1 | 0
  Atrial fibrillation / postoperative period | 8 | 4 | 9
  Atrial flutter / postoperative period | 4 | 0 | 0
Statistical Analysis 1: Comparison: Group 0. vs Group 1 vs Group 2; Hydrothorax / postoperative period; Test type: Superiority; p = 0.6, Chi-squared
Statistical Analysis 2: Comparison: Group 0. vs Group 1 vs Group 2; Hydropericardium / postoperative period; Test type: Superiority; p = 0.2, Chi-squared
Statistical Analysis 3: Comparison: Group 0. vs Group 1 vs Group 2; Resternotomy / postoperative period; Test type: Superiority; p = 0.6, Chi-squared
Statistical Analysis 4: Comparison: Group 0. vs Group 1 vs Group 2; Atrial fibrillation / postoperative period; Test type: Superiority; p = 0.06, Chi-squared
Statistical Analysis 5: Comparison: Group 0. vs Group 1 vs Group 2; Atrial flutter / postoperative period; Test type: Superiority; p = 0.06, Chi-squared

14. Primary Outcome: Left Ventricular Ejection Fraction - Echocardiography - Assessment of Myocardial Contractility on Days 7-14 After Surgical Treatment. Additional Estimation of Safety.
Description: Evaluation of myocardial contractility according to echocardiography, in particular the left ventricular ejection fraction, was carried out within 7-14 days of the postoperative period, depending on the patient's clinical condition, as well as the maximum degree of information content of this study. The lower the indicator, the worse the prognosis of an unfavorable outcome.
Time Frame: 7-14 days of the postoperative period
Population: all patients included in the study
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
percent | 62.1 (1.6) | 56.4 (2.0) | 55.9 (2.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.4, RepeatedMeasures ANOVA

15. Primary Outcome: Assessment of Myocardial Contractility on Days 7-14 After Surgical Treatment - Echocardiography (Size of the Left Ventricle - Index). Additional Estimation of Safety.
Description: Assessment of myocardial contractility according to echocardiography, in particular the size of the left ventricle - its index, was carried out within 7-14 days of the postoperative period, depending on the clinical condition of the patient, as well as on the maximum information content of this study. The higher the indicator (left ventricular size - index), the worse the prognosis of an unfavorable outcome.
  The index is used as an indicator of payment to obtain a more reliable result (taking into account the individual characteristics of each patient).
  index - left ventricular size (mm.)/ body mass index (kg/m^2).
Time Frame: 7-14 days after surgery
Population: All patients included in the study.
Measure: Mean (Standard Deviation); unit: mm/m^2
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mm/m^2
  Lvd ind. | 2.6 (0.08) | 3 (0.1) | 2.7 (0.1)
  Lvs ind. | 1.8 (0.07) | 2.1 (0.09) | 1.9 (0.09)
  LAind. | 2 (0.06) | 2.2 (0.07) | 2.1 (0.08)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Lvd ind. (Lvd mm./BSA kg / cm) - Evaluation of the left ventricular end-diastolic size index; Test type: Superiority; p = 0.5, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Lvs ind. (Lvs mm./BSA kg / cm) - Evaluation of the left ventricular end-systolic size index; Test type: Superiority; p = 0.5, RepeatedMeasures ANOVA
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; LAind. (LA mm./BSA kg / cm) - Left Atrial Size Index Assessment; Test type: Superiority; p = 0.6, RepeatedMeasures ANOVA

16. Primary Outcome: Volume of the Left Ventricle - Index - Echocardiography. Assessment of Myocardial Contractility on Days 7-14 After Surgical Treatment. Additional Estimation of Safety.
Description: Evaluation of myocardial contractility according to echocardiography, in particular volume of the left ventricle - index was carried out within 7-14 days of the postoperative period, depending on the patient's clinical condition, as well as the maximum degree of information content of this study. The greater the figure (volume of the left ventricle - index), the worse the prognosis of adverse outcome.
  The index is used as an indicator of the payment to obtain a more reliable result (taking into account individual characteristics of each patient).
  index - volume of the left ventricle (ml.)/ body mass index (kg / m^2).
Time Frame: 7-14 days after surgery
Population: All patients included in the study
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mL/m^2
  LVEDV MOD BP ind | 58.8 (4.8) | 70.9 (6.9) | 63.9 (5.9)
  LVESV MOD BP ind. | 23.5 (3) | 31.9 (4.4) | 27.8 (3.7)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; LVEDV MOD BP ind. (LVEDV MOD BP ml./BSA kg / cm) - Evaluation of the left ventricular end-diastolic volume index; Test type: Superiority; p = 0.4, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Evaluation of the left ventricular end-systolic volume index (LVESV MOD BP ind.); Test type: Superiority; p = 0.3, RepeatedMeasures ANOVA

17. Primary Outcome: Restoration of the Heart Rate After the Completion of the Main Stage of the Surgical Intervention. Additional Estimation of Safety.
Description: The need to perform defibrillation to restore sinus rhythm, at the end of the main stage of surgery.
Time Frame: Upon completion of the main stage of surgery.
Population: All patients included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
Participants | 3 | 3 | 4
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.6, Chi-squared

18. Secondary Outcome: All-cause Mortality Associated With the Progression of Basic Disease.
Description: The total number of deaths - in the primary hospitalization and during the observation period of 12 months after surgical treatment - deaths associated with the progression of the initial disease.
  The complication rate for CABG operations is 30±10%. According to n1=kn2; n1 sample size, in the control. In group 0, k=2/3 times more than in group 1 and group 2. The difference between the test and control frequencies is ε=p1-p2. Accordingly, with p1 = 0.2; p2=0.4, δ= 0.1; n1=49.5, n2=33. The result is group 0 - 36, group 1 and 2 - 25+25 = 50. The null hypothesis of complication rate δ.All patients included in the study.
Time Frame: 12 months after surgery
Population: All patients included in the study (groups 1 and 2) were compared with the control group (Group 0).In patients included in study during the observation period after the treatment there was no progression of the underlying disease that was fatal.
Measure: Number; unit: participants
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
participants | 0 | 0 | 0

19. Secondary Outcome: Quality of Life. Evaluation of the Quality of Life (Minnesota Questionnaire (MHFLQ), Seattle Questionnaire (SAQ), SF-36 Questionnaire). Estimation of Efficiency.
Description: The SF-36 questionnaire. The indicators of each scale vary between 0 and 100, where 100 represents total health. The results are presented in the form of scores on 8 scales, compiled in such a way that a higher score indicates a higher level of quality of life.MHFLQ - for patients with heart failure.The specified questionnaire consists of 21 questions. To answer each question, a scale of 6 points from the minimum intensity of certain symptoms to the maximum is used. The assessment is based on the sum of points, where the maximum number of points - 105 corresponds to the patient's worst condition. The lowest score 0 points is the best clinical condition of the patient. SAQ consists of 19 questions about the patient's condition, which are divided into the following 5 scales. The quality of life for each of the five scales under consideration is measured in percent, with 0% corresponding to the worst quality of life, and 100% to the best.
Time Frame: At baseline and after one year.
Population: All patients included in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
score on a scale
  Physical Functioning SF-36 | 48.6 (4.6) | 47.8 (6.2) | 51.1 (6.2)
  Physical Functioning SF-36 in year | 62.9 (4) | 69.2 (5.4) | 68.6 (5.4)
  Role-Physical Functioning SF-36 | 24.2 (6.2) | 20.8 (8.4) | 21 (8.4)
  Role-Physical Functioning SF-36 in year | 38.7 (7.4) | 41.7 (10) | 43.06 (10)
  Bodily pain SF-36 | 50.9 (4.9) | 53.3 (6.7) | 57.8 (6.7)
  Bodily pain SF-36 in year | 68 (4.5) | 75.8 (6.04) | 73.4 (6.04)
  General Health SF-36 | 48.6 (2.5) | 50.1 (3.4) | 45 (3.4)
  General Health SF-36 in year | 52.4 (2.4) | 53.2 (3.3) | 53.5 (3.3)
  Vitality SF-36 | 52.6 (3.7) | 54.7 (4.9) | 53.8 (4.9)
  Vitality SF-36 in year | 61.3 (2.6) | 67.2 (3.6) | 64.7 (3.6)
  Social Functioning SF-36 | 66.4 (4.2) | 65.9 (5.7) | 66.3 (5.7)
  Social Functioning SF-36 in year | 77.8 (3.9) | 77.08 (5.2) | 82.6 (5.2)
  Role- Emotional SF-36 | 51.5 (7.2) | 40.7 (9.7) | 38.3 (9.7)
  Role- Emotional SF-36 in year | 58.6 (7.6) | 53.7 (10.2) | 55.5 (10.2)
  Mental Health SF-36 | 60.6 (3.1) | 64.9 (4.2) | 67.5 (4.2)
  Mental Health SF-36 in year | 64.5 (2.9) | 70 (3.98) | 72.7 (3.98)
  Minnesota Quality of Life (MHFLQ) | 39.8 (3.6) | 35.1 (4.9) | 33.3 (4.9)
  Minnesota Quality of Life (MHFLQ) in year | 31.6 (2.9) | 22.7 (3.9) | 22.1 (3.9)
  Seattle QuestionnairePhysical limitation | 39.6 (3.5) | 42.6 (5.4) | 40 (5.2)
  SeattleQuestionnairePhysical limitation / in year | 53.5 (2.9) | 60.8 (4.4) | 58.6 (4.3)
  SeattleQuestionnaireAngina stability | 43.5 (6.3) | 40.4 (9.7) | 61 (9.4)
  SeattleQuestionnaireAngina stability / in year | 87 (7.1) | 91.9 (10.9) | 98.2 (10.6)
  SeattleQuestionnaireAngina frequency | 48.7 (5.7) | 48.5 (8.8) | 46.07 (8.5)
  SeattleQuestionnaiAngina frequency / in year | 80.3 (4.2) | 90.8 (6.6) | 86.4 (6.3)
  SeattleQuestionnaireTreatment satisfaction | 58.9 (3.7) | 72.1 (5.8) | 69.6 (5.6)
  SeattleQuestionnaireTreatmentSatisfaction/ in year | 75.2 (3.2) | 81.3 (4.9) | 80.4 (4.8)
  SeattleQuestionnaire Disease perception | 41.4 (4.3) | 36.5 (6.7) | 37.9 (6.5)
  SeattleQuestionnaire Disease perception/ in year | 60.7 (24.4) | 64.2 (20.8) | 64.3 (20.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Physical Functioning SF-36. Comparison of patients of group 1 and group 2 with the control group - group 0; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Role-Physical Functioning SF-36; Test type: Superiority; p = 0.8, RepeatedMeasures ANOVA
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; Bodily pain SF-36; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 4: Comparison: Group 0 vs Group 1 vs Group 2; General Health SF-36; Test type: Superiority; p = 0.6, RepeatedMeasures ANOVA
Statistical Analysis 5: Comparison: Group 0 vs Group 1 vs Group 2; Vitality SF-36; Test type: Superiority; p = 0.8, RepeatedMeasures ANOVA
Statistical Analysis 6: Comparison: Group 0 vs Group 1 vs Group 2; Social Functioning SF-36; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 7: Comparison: Group 0 vs Group 1 vs Group 2; Role- Emotional SF-36; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 8: Comparison: Group 0 vs Group 1 vs Group 2; Mental Health SF-36; Test type: Superiority; p = 0.96, RepeatedMeasures ANOVA
Statistical Analysis 9: Comparison: Group 0 vs Group 1 vs Group 2; Minnesota Quality of Life (MHFLQ); Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 10: Comparison: Group 0 vs Group 1 vs Group 2; Seattle QuestionnairePhysical limitation; Test type: Superiority; p = 0.6, RepeatedMeasures ANOVA
Statistical Analysis 11: Comparison: Group 0 vs Group 1 vs Group 2; SeattleQuestionnaireAngina stability; Test type: Superiority; p = 0.4, RepeatedMeasures ANOVA
Statistical Analysis 12: Comparison: Group 0 vs Group 1 vs Group 2; SeattleQuestionnaireAngina frequency; Test type: Superiority; p = 0.6, RepeatedMeasures ANOVA
Statistical Analysis 13: Comparison: Group 0 vs Group 1 vs Group 2; SeattleQuestionnaireTreatment satisfaction; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA
Statistical Analysis 14: Comparison: Group 0 vs Group 1 vs Group 2; SeattleQuestionnaire Disease perception; Test type: Superiority; p = 0.3, RepeatedMeasures ANOVA

20. Secondary Outcome: Assessment of the Functional Class of Exertional Angina at 12 Months After Surgical Treatment.
Description: 1. functional class - The usual load does not cause changes in the state of health. Painful attacks occur against the background of excessive loads - after climbing several flights of stairs, while walking fast.
  2. functional class - Pain attacks when walking more than 500 meters, when climbing stairs more than one floor.
  3. functional class - The patient does not tolerate minimal physical activity. An attack occurs when walking a distance of 50-100 meters. Climbing stairs is difficult.
  4. functional class - Activity is significantly limited. Angina pectoris manifests itself when performing minimal actions, including at rest.
Time Frame: up to 12 months
Population: Data analysis of all patients underwent follow-up examination 12 months after surgery.
Measure: Number; unit: participants
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
participants
  1 functional class of angina pectoris1 year after | 15 | 4 | 5
  2 functional class of angina pectoris1 year after | 7 | 0 | 0
  3 functional class of angina pectoris1 year after | 0 | 0 | 0
  4 functional class of angina pectoris1 year after | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.001, Chi-squared

21. Secondary Outcome: Dynamics of the Functional Class of Heart Failure (NYHA). Estimation of Efficiency.
Description: 1. functional class - There is no limitation of a person's physical activity, shortness of breath manifests itself when going above the third floor.
  2. functional class - slight limitation of activity, palpitations, shortness of breath, fatigue occur during normal physical activity and more.
  3. functional class - Symptoms occur with the smallest physical activity, resulting in a significant decrease in activity. At rest, clinical manifestations are not observed.
  The smaller the functional class, the better the quality of human life.
Time Frame: Assessment of the dynamics at 12 months after treatment.
Population: In one case, a patient of Groups 1 through 12 months after the treatment, marked progression of the functional class of heart failure. It should be noted that this patient did not adhere to the recommendations on lifestyle and drug therapy in the postoperative period.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Coronary artery bypass grafting with intramyocardial administration of autologous bone marrow stem cells 0.2 ml - 10 injection in the zone of blood supply LAD.
- Group 2: Coronary artery bypass grafting with intramyocardial (0.2 ml - 10 injection in the zone of blood supply LAD) and intracoronary administration of autologous bone marrow stem cells.
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
Participants
  1 functional class heart failure (NYHA). | 12 | 14 | 7
  2 functional class heart failure (NYHA). | 25 | 10 | 15
  3 functional class heart failure (NYHA). | 0 | 1 | 0
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.13, Chi-squared

22. Secondary Outcome: Evaluation of the Left Ventricular Ejection Fraction 12 Months After Treatment.
Description: According to echocardiography.
Time Frame: 12 months after treatment.
Population: All patients included in the study.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
percent | 61.4 (1.5) | 58.1 (1.8) | 58.4 (1.9)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.35, RepeatedMeasures ANOVA

23. Secondary Outcome: Estimation of the Index of Linear Parameters of the Left Ventricle 12 Months After the Treatment. Estimation of Efficiency.
Description: Evaluation of myocardial contractility according to echocardiography, in particular the size of the left ventricle - the index was carried out 12 months after CABG. The higher the indicator (left ventricular size - index), the worse the prognosis of an unfavorable outcome.
  The index is used as an indicator of the payment to obtain a more reliable result (taking into account individual characteristics of each patient).
  index - size of the left ventricle (mm.)/ body mass index (kg/m^2).
Time Frame: 12 months after the treatment.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: mm/m^2
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mm/m^2
  Lvd ind. | 2.7 (0.07) | 2.9 (0.08) | 2.8 (0.09)
  Lvs ind. | 1.9 (0.06) | 2.07 (0.08) | 1.8 (0.08)
  LAind. | 2.2 (0.05) | 2.3 (0.07) | 2.2 (0.07)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Lvd ind. (Lvd mm./BSA) - left ventricular end-diastolic size index. All patients included in the study; Test type: Superiority; p = 0.2, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Lvs ind. (Lvs mm./BSA kg / cm) - left ventricular end-systolic size index; Test type: Superiority; p = 0.2, RepeatedMeasures ANOVA
Statistical Analysis 3: Comparison: Group 0 vs Group 1 vs Group 2; LAind. (LA mm./BSA kg / cm) - left atrial index; Test type: Superiority; p = 0.5, RepeatedMeasures ANOVA

24. Secondary Outcome: Estimation of the Index of Volumetric Parameters of the Left Ventricle 12 Months After the Treatment. Estimation of Efficiency.
Description: Evaluation of myocardial contractility according to echocardiography, in particular the volume of the left ventricle - the index was carried out 12 months after CABG. The higher the indicator (left ventricular volume - index), the worse the prognosis of an unfavorable outcome.
  The index is used as an indicator of the payment to obtain a more reliable result (taking into account individual characteristics of each patient).
  index - volume of the left ventricle (mm.)/ body mass index (kg/m^2).
Time Frame: 12 Months After the Treatment
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
mL/m^2
  LVEDV MOD BP ind. | 62.3 (4.4) | 70.4 (6.2) | 66.9 (5.5)
  LVESV MOD BP ind. | 25.2 (2.6) | 31.5 (3.9) | 25.6 (3.5)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; LVEDV MOD BP ind. (LVEDV MOD BP ml./BSA kg / cm) - left ventricular end-diastolic volume index; Test type: Superiority; p = 0.6, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; LVESV MOD BP ind. (LVESV MOD BP ml./BSA kg / cm) - left ventricular end-systolic volume index; Test type: Superiority; p = 0.2, RepeatedMeasures ANOVA

25. Secondary Outcome: Assessment of Left Ventricular Diastolic Function - Peak E of Transmitral Flow and Peak А of Transmitral Flow 12 Months After Treatment.
Description: Evaluation of left ventricular diastolic function (echocardiography). The peak velocity E reflects the pressure gradient between the LA and LV in early diastole, and it is affected by preload and disturbance LV relaxation The speed of peak A, which forms at the end diastole, influences LV compliance and contractility left atrium.
Time Frame: 12 months after treatment.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: meters/sec.
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
meters/sec.
  Peak E of transmitral flow | 0.7 (0.04) | 0.7 (0.05) | 0.8 (0.05)
  Peak А of transmitral flow | 0.7 (0.09) | 07 (0.1) | 0.8 (0.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Peak E of transmitral flow; Test type: Superiority; p = 0.35, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; Peak A of transmitral flow; Test type: Superiority; p = 0.7, RepeatedMeasures ANOVA

26. Secondary Outcome: Assessment of Left Ventricular Diastolic Function E/A - 12 Months After Treatment.
Description: The ratio of the transmitral flow, wave E (ejection wave / left ventricular contraction) to wave A (ejection wave / left atrial contraction). The norm is 0.75-1.5 Less than 0.75 violation of relaxation, more than 1.5 restrictive type of diastolic dysfunction.
Time Frame: 12 months after treatment
Population: All patients included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
ratio | 1 (0.1) | 1.2 (0.1) | 1.2 (0.1)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Peak E of transmitral flow/ Peak A of transmitral flow (E/A); Test type: Superiority; p = 0.5, RepeatedMeasures ANOVA

27. Secondary Outcome: Assessment of Left Ventricular Diastolic Function - DT and IVRT 12 Months After Treatment.
Description: Echocardiographic data ( DT (Half-time of wave E), time of isovolumic relaxation of the left ventricle (IVRT).
  DT (Half-time of wave E). The DT time index reflects the relaxation process LV, LV diastolic pressure after mitral valve opening, and LV compliance. 150-200 ms - normal; > 200 ms - violation of relaxation; 150-200 ms - pseudonormal type of left ventricular filling; <150 ms - restrictive type of diastolic dysfunction IVRT (time of isovolumic relaxation of the left ventricl.) <100 ms - normal; > 100 ms - violation of relaxation
Time Frame: 12 Months After Treatment.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
ms
  DT (Half-time of wave E). | 250.4 (15.2) | 252.6 (20.08) | 256.6 (18.3)
  time of isovolumic relaxation of the left ventricle (IVRT). | 96.9 (4.1) | 102.4 (5.5) | 99.6 (4.9)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; DT (Half-time of wave E); Test type: Superiority; p = 0.9, RepeatedMeasures ANOVA
Statistical Analysis 2: Comparison: Group 0 vs Group 1 vs Group 2; time of isovolumic relaxation of the left ventricle; Test type: Superiority; p = 0.9, RepeatedMeasures ANOVA

28. Secondary Outcome: Distance Traveled in the 6-minute Walk Test. Test Results With 6 Minute Walk
Description: The dynamic of the number of meters walked according to the 6-minutes walk test (6MWD) in the observation groups.
Time Frame: initially and after 12 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
meters
  Original number of meters. | 315.06 (17.6) | 319.8 (24.5) | 329.9 (25.3)
  Number of meters in 12 months. | 433.54 (20.6) | 524.4 (28.7) | 452.7 (29.7)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Test type: Superiority; p = 0.0367, Kruskal-Wallis

29. Secondary Outcome: The Number of Functioning Grafts 12 Months After CABG. Patency of Grafts Within a Specified Time of Treatment (Angiography).
Description: According to the angiographic study.
Time Frame: up to 12 months
Population: All patients included in the study.
Measure: Number; unit: Number of grafts
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
Number of grafts
  Initial number of grafts | 113 | 79 | 75
  Number of functioning grafts at 12 months | 99 | 76 | 73
  Number of non-functioning grafts after 12 months | 14 | 3 | 2
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Assessment of the functioning of grafts. Patency of grafts within a specified time of treatment (angiography); Test type: Superiority; p = 0.04, Chi-squared

30. Secondary Outcome: Analysis of the Effect of Left Ventricular Diastolic Dysfunction on the Patency of the Grafts.
Description: Echocardiographic data.
Time Frame: up to 12 months
Population: All patients included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intramyocardial Administration 0.9 % NaCl (Sodium Chloride) - Group 0 | Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1 | Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2
Number analyzed (Participants) | 37 | 25 | 23
Participants
  Number of patients with non-functioning grafts | 10 | 1 | 2
  Patients with non-functioning grafts in the presence of LV diastolic dysfunction after 12 months. | 8 | 0 | 1
Statistical Analysis 1: Comparison: Intramyocardial Administration 0.9 % NaCl (Sodium Chloride) - Group 0 vs Intramyocardial Administration Autologous Bone Marrow Stem Cells - Group 1 vs Intramyocardial and Intracoronary Administration Autologous Bone Marrow Stem Cells - Group 2; Test type: Superiority; p = 0.05, Chi-squared

31. Other Pre Specified Outcome: The Volume of Cellular Material (Cytosis).
Description: Dependence and Duration of Positive Clinical Effect on the Amount of Injected Cell Material (cytosis).
Time Frame: Initial data at the time of collection of bone marrow cells.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: *10^8cells/l
Groups:
- Group 1: Сoronary artery bypass grafting with intramyocardial administration of autologous bone marrow mononuclear cells 0.2 ml - 10 injection in the zone of blood supply LAD.
- Group 2: Сoronary artery bypass grafting with intramyocardial ( 0.2 ml - 10 injection in the zone of blood supply LAD) and intracoronary administration of autologous bone marrow mononuclear cells.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 23
*10^8cells/l | 20.3 (8.9) | 20.3 (8.9)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.05, Discriminant Analysis

32. Other Pre Specified Outcome: The Amount of Cell Material (Percentage).
Description: Dependence and duration of positive clinical effect on the amount of injected cell material (Mononuclear fraction %, CD34+ %, CD133+ %).
  Assessment - mononuclear fraction, CD 34 +, CD 133+ according to flow cytometry data.
Time Frame: Initial data at the time of collection of bone marrow cells.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 23
percent
  Mononuclear fraction/ % | 21.04 (2.9) | 20.0 (2.7)
  CD34+/ % | 1.16 (0.22) | 1.18 (0.34)
  CD133+/ % | 0.4 (0.08) | 0.38 (1.14)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Mononuclear fraction %; Test type: Superiority; p = 0.05, Discriminant Analysis; Data were analyzed by 1, 2, and 3 sections according to the study design
Statistical Analysis 2: Comparison: Group 1 vs Group 2; CD34+ %; Test type: Superiority; p = 0.057, Discriminant Analysis; Data were analyzed by 1, 2, and 3 sections according to the study design
Statistical Analysis 3: Comparison: Group 1 vs Group 2; CD133+ %; Test type: Superiority; p = 0.05, Discriminant Analysis

33. Other Pre Specified Outcome: Smoking as a Factor That Negatively Affects the Results of the Test With a 6-minute Walk in Dynamics.
Description: The distance covered (in meters) was compared with the proper value depending on age (years), height (cm), weight (kg), body mass index (BMI). The due values (6MWD (i)) were calculated using the following formulas: For men: 6МWD (i) = 7.57 × height - 5.02 × age - 1.76 × weight - 309 or 6MWD (i) = 1140 - 5.61 × BMI - 6.94 × age. For women:
  6МWD (i) = 2.11 × height - 2.29 × weight - 5.78 × age + 667 Or 6МWD (i) = 1017 - 6.24 × BMI - 5.83 × age. This difference at baseline is reported as distance walked for smokers minus non-smokers.
Time Frame: 12 months after treatment.
Population: The data of all patients initially included in the study were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group 0 | Group 1 | Group 2
Number analyzed (Participants) | 37 | 25 | 23
meters
  diference between smokers and non-smoking participants at baseline | 230.04 (28.7) | 215.3 (31.4) | 224.8 (27.1)
  diference between baseline and1 year after surgery: number analyzed (Participants) | 30 | 23 | 19
  diference between baseline and1 year after surgery | 87.9 (4.9) | 8.5 (2.7) | 62.1 (4.8)
Statistical Analysis 1: Comparison: Group 0 vs Group 1 vs Group 2; Factor analysis - determining the influence of a factor, in this case, smoking, on the deficit in the number of meters passed according to the test with a 6-minute walk; Test type: Superiority; p = 0.046, Factor analysis

ADVERSE EVENTS:
Time Frame: 12 months after treatment
Arm/Group | Group 0 | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/37 | 0/25 | 0/23

LIMITATIONS AND CAVEATS:
No limitations identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes